CLINICAL TRIAL: NCT05019261
Title: Randomized Trial of a Scalable, Interactive Tool to Support Surrogate Decision-makers of Critically Ill Older Adults
Brief Title: Multi-component Family Support Tool Intervention (FST)
Acronym: FST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Duke University (Other); Baystate Medical Center (Other); Oregon Health and Science University (Other); National Institute on Aging (NIA) (NIH); New York City Health and Hospitals Corporation (Other); VA Pittsburgh Healthcare System (U.S. Federal Agency); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Douglas White, Professor of Critical Care Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY20110367; R01AG066731-01 (NIH)
Record Dates: First submitted 2021-07-30; First posted 2021-08-24 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Critical Illness
Keywords: Patient centeredness of care; Psychological Distress; End of Life Care; Critical Illness; Surrogate Decision Making; Goal Concordant Care
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Multi-component Family Support Intervention
  Interventions: Other: Multi-component Family Support Intervention
- Control (No Intervention): Usual ICU care

INTERVENTIONS:
Other: Multi-component Family Support Intervention — The multi-component intervention is designed to enhance the quality of clinician-family communication and help families manage the emotional and cognitive complexities of surrogate decision-making. It involves: 1) proactive clinician-family meetings; 2) use by surrogates of an interactive web-based tool throughout the ICU stay which is narrated by family members of ICU patients and includes stories and experiences from other families, self-care strategies, brief videos explaining what to expect during family meetings, a question prompt list, an interactive values clarification exercise, and an explanation of different treatment pathways for critically ill patients. 3. Prior to the proactive family meetings, the ICU team is provided with a summary of the family's main questions/concerns, their prognostic expectations, a summary of the patient's values and preferences, and surrogates' current ratings of the extent to which their psychosocial needs are being addressed in the ICU.
  Arms: Intervention

SUMMARY:
The National Academy of Medicine and the National Institutes of Health have called for urgent action to improve the care delivered to the nearly 1,000,000 older Americans who die in intensive care units (ICUs) annually or survive with substantial impairments. These patients often die with distressing symptoms and may receive more invasive, life-prolonging treatment than they would choose for themselves. Moreover, their family members acting as surrogate decision-makers often experience lasting psychological distress from the ICU experience. We will conduct a multicenter randomized trial among 370 incapacitated, critically ill older adult patients at high risk of death or severe functional impairment, their surrogate decision-makers, and their ICU clinicians to determine whether a multi-component family support intervention can improve the patient- and family-centeredness of care (primary outcome), as well as positively impact a variety of other patient, family, and healthcare delivery outcomes. The multicomponent intervention involves: Proactive family meetings scheduled within 48 hours of ICU admission and approximately every 5-7 days after that.

Surrogates will have access (computer, tablet, or mobile phone) to the interactive web-based Family Support Tool. The tool will familiarize families with the ICU and prepare them for their interactions with the clinical team by completing specific sections of the Family Support Tool upon study enrollment, before family meetings, and any other time they wish. The ICU team will receive a tool-generated summary of information about the family before each family meeting, including their main questions and concerns, information about the patient's values and preferences, prognostic expectations, and unmet psychological needs.

DETAILED DESCRIPTION:
The Family Support Tool intervention is designed to help families navigate the emotional, psychological, and cognitive complexities of being a surrogate for an incapacitated critically ill patient and also to enhance the timeliness and quality of clinician-family communication. The intervention consists of three components:

1. Proactive clinician-family meetings within 48 hours of enrollment and every 5-7 days thereafter.
2. Family members complete sections of an interactive web-based tool upon study enrollment, before family meetings, and any other time they wish. Family members can access the tool anywhere via computer, tablet, or mobile phone. The first section of the tool is completed on the first day of study enrollment and contains: video messages supporting families including stories from other families and their experiences and coping strategies, tips on self-care and links to hospital resources. The second and third sections of the FST are completed before scheduled clinician-family meetings on study day 2-3 and again 5-7 days later. These sections of the tool contain: videos detailing what to expect during family meetings, interactive exercises and prompts about patient values, prognosis, care expectations and treatment leanings to help prepare for family meetings. The study team will provide families a printed summary sheet of their main questions for the ICU team that they are encouraged to bring to the family meeting.
3. Before each scheduled family meeting the ICU team receives a written report that summarizes the family's main questions and concerns, information about the patient's values and preferences, surrogates' prognostic expectations, and a visual display of their unmet PC needs.

ELIGIBILITY:
INCLUSION

Patient

1. Age ≥18
2. Lack of decision-making capacity as determined by clinical examination by the attending physician or designee
3. Clinical indication of at least 40% risk of death or ≥40% chance of new, severe long-term functional impairment (needs assistance with ≥ 2 ADLs), as judged by the patient's attending physician or designee

Surrogate

1. The primary surrogate is determined by the patient's advance directive or, if no directive exists, by following the hierarchy of surrogates codified in state law.
2. Up to 3 additional surrogates

Clinician

1. Patient's primary attending (or their designee)

EXCLUSION

Patient

1. Lack of a surrogate decision maker
2. Family not available for study
3. Imminent death (within 24 hours); goals of care are already "comfort measures only"; decision to withdraw life support has already been made
4. Currently participating in a competing research study that does not allow co-enrollment
5. Incarcerated or on an involuntary hold
6. Died prior to enrollment
7. Discharged prior to enrollment
8. Regained capacity prior to enrollment
9. Physician declined patient's participation
10. Physician and designee declined own participation
11. Patient does not meet inclusion criteria within 5 days of ICU admission
12. MD expects transfer orders will be written or the patient will be transferred within 36 hours of screening
13. Greater than 5 ICU days during the current hospitalization

Surrogate

1. Age <18 years
2. Cannot read or understand English
3. Cannot complete questionnaires due to physical or cognitive limitations
4. Has no access to or cannot travel to access the internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1163 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Patient and family centeredness of care | 3 months after hospital discharge
  12-item Patient Perceived Patient-Centeredness of Care Scale (PPPC), previously modified for use by surrogates, completed at 3-month telephone follow-up of surrogates.

SECONDARY OUTCOMES:
Composite measure of goal-concordant care | 3 months after hospital discharge
  Assessed by surrogates at 3-month telephone follow-up using an 8-item composite measure of goal-concordant care.
Satisfaction with ICU care | 3 months after hospital discharge
  Assessed using the Family Satisfaction in the ICU (FS-ICU) instrument at 3-month telephone follow-up of surrogates. The FS-ICU is a 24-item scale concerning satisfaction with care, communication, and decision-making in the ICU.
Unmet palliative care needs | Measured at day 5 post-randomization
  Measured using the adapted Needs of Social Nature, Existential Concerns, Symptoms, and Therapeutic Interaction (NEST) scale administered to surrogates on day 5 post-randomization. The adapted NEST scale is designed for ICU use; it is a 13-item instrument developed to identify unmet social, emotional, physical, and care-system needs in serious illness.
Surrogates' prognostic awareness | Measured at day 5 post-randomization
  Assessed on study day 5 using the validated Clinician-Surrogate Concordance Scale (CSCS), which our research team developed. The single item CSCS has excellent test-retest reliability (r =0.91). It has established criterion validity and responsiveness to change.
Surrogates' clarity about patient values and preferences | Measured at day 5 post-randomization
  Assessed by surrogates after family meetings on study day 5 using the "informed" and "values clarity" subscales, 6 items out of the 16-item Decisional Conflict Scale (DCS). The scale has established responsiveness to change, test-retest reliability (r=0.81), internal consistency (α=0.92), and discriminant validity.
Clinician-family conflict | Measured at day 5 post-randomization
  A brief survey (measured by both surrogates and ICU clinicians) to determine the level of family-clinician conflict during index hospitalization
Perceived effectiveness of Family Support Tool | Measured at day 5 post-randomization
  A brief survey asking (intervention only) surrogate participants perceived effectiveness of the FST intervention
Risk of post-traumatic stress disorder | 6 months after hospital discharge
  Assessed using the Impact of Events Scale-revised (IES-R) at 6 months. The IES-R is a valid, reliable, and responsive 22 -item instrument measuring symptoms of avoidance and intrusive thoughts. A score 33 indicates a high risk of PTSD. It has been used successfully among ICU surrogates.
Surrogates' symptoms of anxiety and depression | 6 months after hospital discharge
  The HADS is a 14-item, two-domain (anxiety, depression) instrument with established reliability and validity among ICU surrogates that is recommended by consensus guidelines for use among ICU surrogates. Assessed at 6-month telephone follow-up.
Resource utilization | 3 months and 6 months after hospital discharge
  Among hospital survivors we will perform interviews with surrogates at 3-months and 6-months to identify patient's post-discharge healthcare utilization (e.g. hospital admissions, ED visits, skilled-nursing facility use, hospice use, etc.), assigning costs using validated methods.
Proportion of patients with new DNR order during index hospitalization and time to first DNR order during index hospitalization | 6 months after hospital discharge
Proportion of patients who received comfort-focused care during the index hospitalization and time to comfort-focused care | 6 months after hospital discharge
Proportion of patients enrolled in hospice during index hospitalization | 6 months after hospital discharge
ICU and hospital length of stay | 6 months after hospital discharge
  Duration of time patient spent in ICU and hospital
Duration of mechanical ventilation | 6 months after hospital discharge
  Duration of time patient spent on mechanical ventilation during index hospitalization
Cost of index hospitalization | 6 months after hospital discharge
  Assigning costs using validated methods, the cost of index hospitalization will be calculated
Time to hospice | 6 months after hospital discharge
  time in days from enrollment to hospice

OTHER OUTCOMES:
Patient hospital survival | 6 months after hospital discharge
  The vital status of the patient will be assessed at the conclusion of index hospitalization
Duration of survival from hospital discharge through 6-month follow-up | 6 months after hospital discharge
  This will be measured as a time-to-event variable, with time 0 being the date of hospital discharge. All death dates will be confirmed by querying the SSDMF or institutional death indices at the completion of the trial.
Days alive outside healthcare facilities | 6 months after hospital discharge
  We will calculate the number of days a patient was alive from discharge to 6 months, then subtract that from the number of days the patient was in a hospital, LTAC, SNF, rehab facility, or hospice.
Patients' functional status | 6 months after hospital discharge
  Assessed using the Katz Index of Independence in Activities of Daily Living, a validated and widely-used scale to quantify patients' functional status. Katz is a 6-item (1 or 0 point) scale measuring independency in older adults. Lower scores indicate a greater level of dependence for measured skills.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas B White, MD, MAS, Principal Investigator — University of Pittsburgh
Locations (7):
- United States (7):
  - Baystate Medical Center, Springfield, Massachusetts
  - NYC Health + Hospitals/Lincoln Hospital, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Pittsburgh VA Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Raw data and derived datasets will be made available to external investigators and the public on a case-by-case basis, to be approved by the PI and in accordance with institutional, HIPAA, state and federal regulations. A data-sharing agreement may be instituted, depending upon the data to be shared. All data that is shared will be de-identified to protect participant privacy and confidentiality. Data and datasets will be retained and available to share for at least three years following completion of the project, in accordance with NIH regulations.